CLINICAL TRIAL: NCT04218617
Title: Single- vs. Two-Fraction Spine Stereotactic Radiosurgery for the Treatment of Vertebral Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE3319
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Spine Metastases; Spine Stereotactic Radiosurgery (sSRS)
Keywords: C79.40; C79.49; C79.51; C79.52

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm 1 - Single fraction (Experimental): sSRS 18 Gy in 1 fraction
  Interventions: Device: Diagnostic MRI; Device: Planning MRI; Other: Simulation CT; Other: QOL assessment; Other: Brief pain inventory (BPI); Radiation: sSRS in 1 fraction
- Arm 2 - Two fraction (Active Comparator): sSRS 24 Gy in 2 fractions
  Interventions: Device: Diagnostic MRI; Device: Planning MRI; Other: Simulation CT; Other: QOL assessment; Other: Brief pain inventory (BPI); Radiation: sSRS in 2 fraction

INTERVENTIONS:
Device: Diagnostic MRI — Diagnostic MRI
Device: Planning MRI — Planning MRI: high definition (HD) MRI of the region of interest (1 vertebral level above and below the level(s) being treated)
Other: Simulation CT — Simulation CT is obtained (1.5 mm slice thickness)
Other: QOL assessment — QOL assessment
Other: Brief pain inventory (BPI) — Brief pain inventory (BPI), including narcotic assessment
Radiation: sSRS in 1 fraction — sSRS 18 Gy in 1 fraction
  Arms: Arm 1 - Single fraction
Radiation: sSRS in 2 fraction — sSRS 24 Gy in 2 fractions to be delivered either on consecutive days or one day apart.
  Arms: Arm 2 - Two fraction

SUMMARY:
Spine radiosurgery (SRS) utilizes advanced treatment planning with focused x-rays to deliver one to four high dose treatments to the spine to help relieve pain and/or neurologic symptoms. Spine SRS uses special equipment to position the participant and guide the focused beams toward the area to be treated and away from normal tissue.

One of the side effects of spine SRS is the development of vertebral compression fractures, many of which are not painful. The goal of this study is to compare the effects, good and/or bad, of spine SRS given in 1 or 2 treatments. Our main goal is to find out which approach will reduce the chances of developing vertebral compression fractures.

DETAILED DESCRIPTION:
The primary objective of this study is to establish the non-inferiority in vertebral compression fracture (VCF) incidence at 6 months between single-fraction and two-fraction sSRS.

Other objectives are to to evaluate the 12-month impact of single- and two-fraction sSRS on local control (LC), pain control (PC), quality of life (QOL), and toxicity (specifically, pain flare, radiation esophagitis/laryngitis/pharyngitis, and radiation myelitis)

This study is planned as a two-arm randomized phase II trial to establish non-inferiority of single fraction sSRS compared to two-fraction sSRS. Approximately 130 participants will be enrolled in this trial; 65 participants in each arm:

* Group 1: If you are assigned to this group, you will undergo spine radiosurgery in a single (1) session.
* Group 2: If you are assigned to this group, you will undergo spine radiosurgery in two (2) sessions.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky Performance Status (KPS) ≥ 70
* RPA class 1 (KPS >70 AND controlled systemic disease) or RPA Class 2 (KPS >70, uncontrolled systemic disease OR KPS ≤70, age ≥54, no visceral metastases)44 (see Appendix II)
* Vertebral metastases from C3 to L5 based on bone scan, CT, PET, or MRI.
* Vertebral metastases must be (1) solitary, (2) at two contiguous levels, or (3) a maximum of three separate sites, with a maximum of two contiguous levels.
* Radioresistant metastases are permitted (including sarcomas, melanomas, and renal cell carcinomas).
* Patients with epidural disease are permitted so long as there is no cord compression.
* Paraspinal extension is permitted, so long as the paraspinal component is ≤5 cm
* Multiple small metastatic lesions (<20% vertebral body involvement) of no clinical correlate are permitted, and not included in the irradiated segments as per RTOG 0631
* History and physical within four weeks of registration.
* Negative pregnancy test within four weeks of registration for women of childbearing potential.
* Diagnostic spine MRI with and without contrast within four weeks of registration
* Neurological exam within four weeks of registration to rule out rapid neurological decline. Mild to moderate neurological deficits are acceptable, as long as distance between lesion and spinal cord is ≥3 mm
* Patients may have prior EBRT at the index site.
* Informed consent of the participant.

Exclusion Criteria:

* Lesions at C1-2 or S1-Coccyx.
* Hematologic malignancies including lymphoma and myeloma.
* Multiple primary cancers.
* Primary neoplasms of the spine
* Prior corpectomy, kyphoplasty/vertebroplasty, or instrumentation at the site of planned sSRS.
* Spinal cord compression.
* Paraspinal mass >5 cm.
* Patients with rapid neurologic decline.
* Bony retropulsion resulting in neurologic deficit.
* Patients with contraindications to MRI.
* Patients allergic to intravenous contrast for MRI or CT.
* Patients with emergent spinal cord compression.
* Patients with mechanical instability of the spine.
* Patients with active connective tissue disease.
* Patients who previously underwent sSRS to the vertebrae of interest.
* Patients with diffuse or multilevel metastatic spinal disease with >20% involvement of vertebral bodies, defined as involvement of >5 vertebral levels.
* Inability to participate in study activities due to physical or mental limitations.
* Inability or unwillingness to return for all required follow-up visits and imaging.
* Inability to deliver sSRS, either 18 Gy in one fraction, or 24 Gy in two fractions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-02-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
6-month cumulative incidence of Vertebral Compression Fracture (VCF) associated with single- and two-fraction sSRS | At baseline and for each subsequent follow-up MRI (at 1 month, 3 months, 6 months and 12 months after treatment)
  6-month cumulative incidence of Vertebral Compression Fracture (VCF) associated with single- and two-fraction sSRS
  Each treated vertebra will be assessed individually for VCF during radiologic follow-up

SECONDARY OUTCOMES:
Local control (LC) as defined as absence of local progression of disease In the event of disease progression, all cases will be reviewed at the multi-disciplinary spine tumor board for a consensus recommendation | At baseline and for each subsequent follow-up MRI (at 1 month, 3 months, 6 months and 12 months after treatment)
  LC as defined as absence of local progression of disease, which include the following:
  1. Gross unequivocal increase in tumor volume or linear dimension.
  2. Any new or progressive tumor within the epidural space.
  3. Neurologic deterioration attributable to pre-existing epidural disease with equivocal increased epidural disease dimensions on MRI.
Pain control (PC) as assessed by the Brief Pain Inventory (BPI) | At baseline and for each subsequent follow-up MRI (at 1 month, 3 months, 6 months and 12 months after treatment)
  PC at each treated vertebral level assessed by the BPI [9 item questionnaire (range: 0-10), higher scores = worse pain], then defined by RTOG 0631 as follows:
  Complete relief (CR): Pain score of 0 at index site 3 mo post-treatment. CR is requisite of no increase in narcotic analgesics.
  Partial relief (PR): Reduction in BPI of ≥ 3 points at index site, provided other treated lesions have increased in pain score and participant did not require increase in narcotic analgesics for site of interest. Participants needing increase in narcotics for site will not be scored as having PR. Those needing increase in narcotics for a distant site will remain eligible for CR/PR.
  Stable response (SR): Post-treatment pain score same as or within 2 points of baseline score at index site with no increase in narcotic analgesics for site of interest.
  Progressive pain: Post-treatment increase of at least 3 points from baseline pain score at index site or increase in narcotics for site of interest.
Quality of life (QOL) assessed by EORTC QLQ-C30 (with BM22) | At baseline and for each subsequent follow-up MRI (at 1 month, 3 months, 6 months and 12 months after treatment)
  Quality of life as measured by (EORTC QOL-C30) - 30 items that are grouped into five scales functional (physical, social, emotional functioning, cognitive and role), three scales of symptoms (fatigue, pain, nausea and vomiting), a global scale of health / quality of life and a number of related individual items with the symptoms of the disease and its treatment, as well as an item of economic impact. The answers to the items on the scales refer to "last week," except the patient's physical functioning scale whose time frame is the present. These answers obey a Likert format, which ranges from 1 ("Not at all") and 4 ("A lot")
Toxicity as assessed by CTCAE V. 5.0 | At follow-up MRI (1 month, 3 months, 6 months and 12 months after treatment)
  Toxicity as assessed by criteria in the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
  Rates of grade 1-5 toxicities will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Chao, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publication, after de-identification
Time Frame: 1 year after last participant is enrolled. Data will be available for a total of 2 years
Access Criteria: Investigators whose purposed use of the data has been approved by the Cleveland Clinic Independent Review Committee. Data will be provided for individual participant meta-analysis. All requests must be made in writing to Sam Chao, MD (Chaos@ccf.org) or Ehsan Balagamwala (Balagae@ccf.org).